CLINICAL TRIAL: NCT05541913
Title: he Effect of Tele-Nursing Service Provided to Parents of Circumcised Children After Discharge on Parents' Anxiety and Care Satisfaction
Brief Title: The Effect of Tele-Nursing on Parents of Circumcised Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Atiye Erbaş, PhD, Duzce University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DuzceUasiye
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Health Care Utilization; Nursing Caries
Keywords: Health care; Care Satisfaction; Tele nursing; Anxiety; Circumcision
MeSH Terms: conditions — Patient Acceptance of Health Care; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Grup (No Intervention): After acceptance of the child's admission to the ward, parents will be asked to complete the Beck Anxiety Scale. Beck Anxiety Scale and Health Care Satisfaction Scale will be applied to the parents again after the discharge training given routinely in the service. Control grup will be called on the postoperative 4th day after discharge and asked to fill in the Beck Anxiety Scale and Health Care Satisfaction Scale.
- Intervention Grup (Experimental): After the admission of the child in the service, the Beck Anxiety Scale will be applied to measure the anxiety levels of the parents at the first hospitalization. After the routine discharge training in the service, the Beck Anxiety Scale and Health Care Satisfaction Scale will be applied to the parents again. Then, the parents will be called on the 1st postoperative day and training will be provided. On the postoperative 2nd, 3rd and 4th days, counseling will be provided. on the postoperative 4th day Parents will be asked to fill in the Beck Anxiety sScale and Health Care Satisfaction scale.
  Interventions: Other: Tele nursing

INTERVENTIONS:
Other: Tele nursing — The intervention group in the study will be the parents of children who received routine care in the surgical service and who received tele-nursing service, who had undergone circumcision operation.After the admission of the child in the service, the Beck Anxiety Scale will be applied to measure the anxiety levels of the parents at the first hospitalization. After the routine discharge training in the service, the Beck Anxiety Scale and Health Care Satisfaction Scale will be applied to the parents again. Then, the parents will be called on the 1st postoperative day and training will be provided. On the postoperative 2nd, 3rd and 4th days, counseling will be provided. on the postoperative 4th day Parents will be asked to fill in the Beck Anxiety sScale and Health Care Satisfaction scale.
  Arms: Intervention Grup

SUMMARY:
Circumcision is applied in many regions of the world for cultural, social, religious and medical reasons. Considering the frequency of circumcision in the World is 30%, this rate is close to 100% in Turkey.

DETAILED DESCRIPTION:
Circumcision is applied in many regions of the world for cultural, social, religious and medical reasons. Considering the frequency of circumcision in the World is 30%, this rate is close to 100% in Turkey. It will be done to determine the effect of the tele-nursing service applied to the parents of circumcised children after discharge on the anxiety and care satisfaction of the parents.

This study is planned to be carried out in Bursa Kestel State Hospital, Surgery Service, between October 2022 and January 2024. This study will consist of a control and an experiment group. This study is planned to be done as a single blind randomised control trial and will use equal samples block randomisation design. The study is planned to carry out with 84 parents, 42 parents in each group.Samples number is calculated via G-power pogramme.

Control grup: The control group in the study will be the parents of children who received routine care in the surgical service and had circumcision operation.After acceptance of the child's admission to the ward, parents will be asked to complete the Beck Anxiety Scale. Beck Anxiety Scale and Health Care Satisfaction Scale will be applied to the parents again after the discharge training given routinely in the service. Control grup will be called on the postoperative 4th day after discharge and asked to fill in the Beck Anxiety Scale and Health Care Satisfaction Scale.

The intervention group: The intervention group: in the study will be the parents of children who received routine care in the surgical service and tele-nursing service, who had undergone circumcision operation.After the admission of the child in the service, the Beck Anxiety Scale will be applied to measure the anxiety levels of the parents at the first hospitalization. After the routine discharge training in the service, the Beck Anxiety Scale and Health Care Satisfaction Scale will be applied to the parents again. Then, the parents will be called on the 1st postoperative day and training will be provided. On the postoperative 2nd, 3rd and 4th days, counseling will be provided. on the postoperative 4th day Parents will be asked to fill in the Beck Anxiety sScale and Health Care Satisfaction scale.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose children will be circumcised,
* At least one parent as a caregiver during the surgical process,
* Parents who are able to read and write -Parents have no communication problems, -
* Parents who can access a smartphone,

Exclusion Criteria:

* Parents who have a childs with a special condition who has difficulties in understanding and perceiving

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Decreasing Anxiety | received tele-nursing service on the postoperative 4th day
  A decrease in anxiety level of parents who received tele-nursing service compared to those who received normal discharge training
Increasing Health Care Satisfaction | received tele-nursing service on the postoperative 4th day
  An increase in the level of care satisfaction of parents who received tele-nursing service compared to those who received normal discharge training

CONTACTS AND LOCATIONS:
Locations (1):
- Atiye Erbaş, Multiple Locations, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No